CLINICAL TRIAL: NCT01960855
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Investigate the Safety and Efficacy of ABT-494 Given With Methotrexate (MTX) in Subjects With Moderately to Severely Active Rheumatoid Arthritis (RA) Who Have Had an Inadequate Response or Intolerance to Anti-TNF Biologic Therapy
Brief Title: A Study Investigating the Efficacy and Safety of ABT-494 Given With Methotrexate in Subjects With Rheumatoid Arthritis Who Failed Anti-Tumor Necrosis Factor (TNF) Biologic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-550; 2013-002358-57 (EudraCT Number)
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis
Keywords: anti-inflammatory agents; Joint Diseases; Arthritis; Musculoskeletal Disease; antirheumatic agents
MeSH Terms: conditions — Arthritis, Rheumatoid; Joint Diseases; Arthritis; Musculoskeletal Diseases | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (5):
- Placebo BID (Placebo Comparator): Placebo twice daily (BID) for 12 weeks.
  Interventions: Drug: Placebo
- ABT-494 3 mg BID (Experimental): ABT-494 3 mg twice daily (BID) for 12 weeks.
  Interventions: Drug: ABT-494
- ABT-494 6 mg BID (Experimental): ABT-494 6 mg twice daily (BID) for 12 weeks.
  Interventions: Drug: ABT-494
- ABT-494 12 mg BID (Experimental): ABT-494 12 mg twice daily (BID) for 12 weeks.
  Interventions: Drug: ABT-494
- ABT-494 18 mg BID (Experimental): ABT-494 18 mg twice daily (BID) for 12 weeks.
  Interventions: Drug: ABT-494

INTERVENTIONS:
Drug: ABT-494 — ABT-494 capsule administered orally twice daily (BID).
  Arms: ABT-494 12 mg BID; ABT-494 18 mg BID; ABT-494 3 mg BID; ABT-494 6 mg BID
Drug: Placebo — Placebo for ABT-494 capsule administered orally twice daily (BID).
  Arms: Placebo BID

SUMMARY:
The primary objective is to compare the safety and efficacy of multiple doses of ABT-494 versus placebo in moderately to severely active RA subjects on stable background MTX therapy with inadequate response or intolerance to anti-TNF biologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis (RA) based on either the 1987-revised American College of Rheumatology (ACR) classification criteria or the 2010 American College of Rheumatology/European League against Rheumatism (ACR/EULAR) criteria for ≥ 3 months.
* Subjects must have been receiving oral or parenteral methotrexate (MTX) therapy ≥ 3 months and on a stable prescription of 7.5 to 25 mg/week for at least 4 weeks prior to initiating the study drug. Subjects should also be on a stable dose of folic acid (or equivalent) for at least 4 weeks prior to initiating the study drug. Subjects should continue with their stable doses of MTX and folic acid throughout the study
* Subjects have been treated with 1 or more anti-tumor necrosis factor (TNF) biologics (no maximum cap) for ≥ 3 months but continue to exhibit active RA, or had to discontinue due to intolerability or toxicity. In addition, subjects with prior exposure to non-anti-TNF biologic(s) (no maximum cap) (e.g., abatacept, rituximab, anakinra, or tocilizumab) are allowed.
* Have active RA as defined by the following minimum disease activity criteria: ≥ 6 swollen joints (based on 66 joint counts) at Screening and Baseline, ≥ 6 tender joints (based on 68 joint counts) at Screening and Baseline, high sensitivity C reactive protein (hs-CRP) > Upper Limit of Normal (ULN) OR positive for both rheumatoid factor and anti-cyclic citrullinated peptide (anti-CCP) antibody.

Exclusion Criteria:

* Prior exposure to Janus Activated Kinase (JAK) inhibitor (e.g. tofacitinib, baricitinib)
* Pregnant or breastfeeding female
* Ongoing or active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kremer JM, Emery P, Camp HS, Friedman A, Wang L, Othman AA, Khan N, Pangan AL, Jungerwirth S, Keystone EC. A Phase IIb Study of ABT-494, a Selective JAK-1 Inhibitor, in Patients With Rheumatoid Arthritis and an Inadequate Response to Anti-Tumor Necrosis Factor Therapy. Arthritis Rheumatol. 2016 Dec;68(12):2867-2877. doi: 10.1002/art.39801. PMID 27389975
- [Derived] Yamaoka K, Tanaka Y, Kameda H, Khan N, Sasaki N, Harigai M, Song Y, Zhang Y, Takeuchi T. The Safety Profile of Upadacitinib in Patients with Rheumatoid Arthritis in Japan. Drug Saf. 2021 Jun;44(6):711-722. doi: 10.1007/s40264-021-01067-x. Epub 2021 May 27. PMID 34041702
- [Derived] Nader A, Mohamed MF, Winzenborg I, Doelger E, Noertersheuser P, Pangan AL, Othman AA. Exposure-Response Analyses of Upadacitinib Efficacy and Safety in Phase II and III Studies to Support Benefit-Risk Assessment in Rheumatoid Arthritis. Clin Pharmacol Ther. 2020 Apr;107(4):994-1003. doi: 10.1002/cpt.1671. Epub 2019 Nov 30. PMID 31610021
- [Derived] Mohamed MF, Klunder B, Camp HS, Othman AA. Exposure-Response Analyses of Upadacitinib Efficacy in Phase II Trials in Rheumatoid Arthritis and Basis for Phase III Dose Selection. Clin Pharmacol Ther. 2019 Dec;106(6):1319-1327. doi: 10.1002/cpt.1543. Epub 2019 Aug 23. PMID 31194885
- [Derived] Klunder B, Mohamed MF, Othman AA. Population Pharmacokinetics of Upadacitinib in Healthy Subjects and Subjects with Rheumatoid Arthritis: Analyses of Phase I and II Clinical Trials. Clin Pharmacokinet. 2018 Aug;57(8):977-988. doi: 10.1007/s40262-017-0605-6. PMID 29076110

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a screening period of 30 days.
Period: Overall Study
Arm/Group | Placebo BID | ABT-494 3 mg BID | ABT-494 6 mg BID | ABT-494 12 mg BID | ABT-494 18 mg BID
Started | 56 | 55 | 55 | 55 | 55
Completed | 45 | 51 | 46 | 51 | 50
Not Completed | 11 | 4 | 9 | 4 | 5
Not completed — Subject noncompliant | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 6 | 2 | 2
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 1 | 1 | 0
Not completed — Consent withdrawn by subject | 3 | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BID | ABT-494 3 mg BID | ABT-494 6 mg BID | ABT-494 12 mg BID | ABT-494 18 mg BID | Total
Number analyzed (Participants) | 56 | 55 | 55 | 55 | 55 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.04) | 57 (13.06) | 56.3 (11.71) | 59.1 (11.4) | 56.7 (12.39) | 57.3 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 43 | 43 | 45 | 42 | 221
  Male | 8 | 12 | 12 | 10 | 13 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: Response defined as at least 20% reduction (improvement) compared with baseline in tender joint count (TJC68), swollen joint count (SJC66), and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, patient's global assessment of disease activity (PtGA); physician's global assessment of disease activity (PGA), Health Assessment Questionnaire - Disability Index (HAQ-DI), and high-sensitivity C-reactive protein (hs CRP). Last observation carried forward (LOCF) was used for missing data.
Time Frame: Baseline (Week 0) and Week 12
Population: Subjects in the modified intent-to-treat (mITT) population with a baseline value and at least 1 post-baseline value
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | ABT-494 3 mg BID | ABT-494 6 mg BID | ABT-494 12 mg BID | ABT-494 18 mg BID
Number analyzed (Participants) | 54 | 54 | 52 | 55 | 55
Participants | 19 | 30 | 33 | 40 | 39
Statistical Analysis 1: Comparison: Placebo BID vs ABT-494 3 mg BID; Test type: Other; p = 0.033, Chi-squared
Statistical Analysis 2: Comparison: Placebo BID vs ABT-494 6 mg BID; Test type: Other; p = 0.004, Chi-squared
Statistical Analysis 3: Comparison: Placebo BID vs ABT-494 12 mg BID; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 4: Comparison: Placebo BID vs ABT-494 18 mg BID; Test type: Other; p < 0.001, Chi-squared

2. Secondary Outcome: Number of Subjects Achieving American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Response defined as at least 50% reduction (improvement) compared with baseline in tender joint count (TJC68), swollen joint count (SJC66), and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, PtGA; PGA, HAQ-DI, and hs CRP. LOCF was used.
Time Frame: Baseline (Week 0) and Week 12
Population: Subjects in the mITT population with a baseline value and at least 1 post-baseline value.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | ABT-494 3 mg BID | ABT-494 6 mg BID | ABT-494 12 mg BID | ABT-494 18 mg BID
Number analyzed (Participants) | 53 | 54 | 52 | 55 | 55
Participants | 9 | 13 | 20 | 24 | 22
Statistical Analysis 1: Comparison: Placebo BID vs ABT-494 3 mg BID; Test type: Other; p = 0.364, Chi-squared
Statistical Analysis 2: Comparison: Placebo BID vs ABT-494 6 mg BID; Test type: Other; p = 0.014, Chi-squared
Statistical Analysis 3: Comparison: Placebo BID vs ABT-494 12 mg BID; Test type: Other; p = 0.003, Chi-squared
Statistical Analysis 4: Comparison: Placebo BID vs ABT-494 18 mg BID; Test type: Other; p = 0.008, Chi-squared

3. Secondary Outcome: Number of Subjects Achieving American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Response defined as at least 70% reduction (improvement) compared with baseline in tender joint count (TJC68), swollen joint count (SJC66), and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, PtGA; PGA, HAQ-DI, and hs CRP. LOCF was used.
Time Frame: Baseline (Week 0) and Week 12
Population: Subjects in the mITT population with a baseline value and at least 1 post-baseline value.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | ABT-494 3 mg BID | ABT-494 6 mg BID | ABT-494 12 mg BID | ABT-494 18 mg BID
Number analyzed (Participants) | 55 | 54 | 52 | 55 | 55
Participants | 2 | 7 | 14 | 12 | 12
Statistical Analysis 1: Comparison: Placebo BID vs ABT-494 3 mg BID; Test type: Other; p = 0.093, Chi-squared
Statistical Analysis 2: Comparison: Placebo BID vs ABT-494 6 mg BID; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Placebo BID vs ABT-494 12 mg BID; Test type: Other; p = 0.004, Chi-squared
Statistical Analysis 4: Comparison: Placebo BID vs ABT-494 18 mg BID; Test type: Other; p = 0.004, Chi-squared

4. Secondary Outcome: Number of Subjects Achieving Low Disease Activity (LDA) Based on Disease Activity Score (DAS28) or Clinical Remission (CR) Based on (DAS28) at Week 12
Description: LDA is defined as DAS28 from 2.6 to < 3.2 at Week 12. CR is defined as DAS28 (CRP) < 2.6 at Week 12. The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, hs CRP, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. LOCF was used.
Time Frame: Baseline (Week 0) and Week 12
Population: Subjects in the mITT population with a baseline value and at least 1 post-baseline value.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | ABT-494 3 mg BID | ABT-494 6 mg BID | ABT-494 12 mg BID | ABT-494 18 mg BID
Number analyzed (Participants) | 55 | 54 | 53 | 55 | 55
Participants | 14 | 18 | 20 | 29 | 25
Statistical Analysis 1: Comparison: Placebo BID vs ABT-494 3 mg BID; Test type: Other; p = 0.366, Chi-squared
Statistical Analysis 2: Comparison: Placebo BID vs ABT-494 6 mg BID; Test type: Other; p = 0.17, Chi-squared
Statistical Analysis 3: Comparison: Placebo BID vs ABT-494 12 mg BID; Test type: Other; p = 0.003, Chi-squared
Statistical Analysis 4: Comparison: Placebo BID vs ABT-494 18 mg BID; Test type: Other; p = 0.028, Chi-squared

5. Secondary Outcome: Number of Subjects Achieving CR Based on DAS28 at Week 12
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, hs CRP, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. LOCF was used.
Time Frame: Baseline (Week 0) and Week 12
Population: Subjects in the mITT population with a baseline value and at least 1 post-baseline value.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | ABT-494 3 mg BID | ABT-494 6 mg BID | ABT-494 12 mg BID | ABT-494 18 mg BID
Number analyzed (Participants) | 55 | 54 | 53 | 55 | 55
Participants | 7 | 13 | 14 | 18 | 17
Statistical Analysis 1: Comparison: Placebo BID vs ABT-494 3 mg BID; Test type: Other; p = 0.126, Chi-squared
Statistical Analysis 2: Comparison: Placebo BID vs ABT-494 6 mg BID; Test type: Other; p = 0.072, Chi-squared
Statistical Analysis 3: Comparison: Placebo BID vs ABT-494 12 mg BID; Test type: Other; p = 0.012, Chi-squared
Statistical Analysis 4: Comparison: Placebo BID vs ABT-494 18 mg BID; Test type: Other; p = 0.021, Chi-squared

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) were collected from first dose of study drug until up to 30 days after discontinuation of study drug (up to 16 weeks); SAEs were collected from the time informed consent was obtained (20 weeks).
Arm/Group | Placebo BID | ABT-494 3 mg BID | ABT-494 6 mg BID | ABT-494 12 mg BID | ABT-494 18 mg BID
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55 | 0/55 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/56 | 2/55 | 2/55 | 0/55 | 1/55
Other Adverse Events (participants affected / at risk) | 9/56 | 13/55 | 9/55 | 14/55 | 27/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo BID (N=56) | ABT-494 3 mg BID (N=55) | ABT-494 6 mg BID (N=55) | ABT-494 12 mg BID (N=55) | ABT-494 18 mg BID (N=55)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo BID (N=56) | ABT-494 3 mg BID (N=55) | ABT-494 6 mg BID (N=55) | ABT-494 12 mg BID (N=55) | ABT-494 18 mg BID (N=55)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (7)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (3) | 4 (4)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
SINUSITIS (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (5) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 7 (9)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (2) | 3 (3) | 3 (4) | 3 (4) | 3 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.